CLINICAL TRIAL: NCT02246439
Title: Randomized, Placebo-Controlled, Phase 3 Trial of BEKINDA (Ondansetron 24 mg Bimodal Release Tablets) for Vomiting Due to Presumed Acute Gastroenteritis or Gastritis (The GUARD Study)
Brief Title: BEKINDA (Ondansetron 24 mg Bimodal Release Tablets) for Vomiting Due to Presumed Acute Gastroenteritis or Gastritis
Acronym: GUARD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: RedHill Biopharma Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RHB-102-01
Record Dates: First submitted 2014-09-16; First posted 2014-09-22 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-01

CONDITIONS: Gastroenteritis; Gastritis
Keywords: Gastroenteritis; Gastritis; Vomiting; Nausea; Diarrhea
MeSH Terms: conditions — Gastroenteritis; Gastritis; Vomiting; Nausea; Diarrhea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- RHB-102 (Experimental): RHB-102, Bimodal Release Ondansetron Tablets
  Interventions: Drug: RHB-102
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: RHB-102 — RHB-102, Bimodal Release Ondansetron Tablets
  Arms: RHB-102
Drug: Placebo Oral Tablet — Placebo
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Randomized, Placebo-Controlled, Phase 3 Trial of RHB-102 (BEKINDA) (Ondansetron 24 mg Bimodal Release Tablets) for Acute Gastroenteritis.

The study will evaluate the safety and efficacy of RHB-102 (BEKINDA) in treating Acute Gastroenteritis, by comparing it to placebo.

DETAILED DESCRIPTION:
Randomized, Placebo-Controlled, Phase 3 Trial of RHB-102 (BEKINDA) (Ondansetron 24 mg Bimodal Release Tablets) for Acute Gastroenteritis.

The study will evaluate the safety and efficacy of RHB-102 (BEKINDA) in treating Acute Gastroenteritis, by comparing it to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have vomited at least twice in the 4 hours preceding signing informed consent. A vomiting episode is defined as an episode of forceful expulsion of stomach contents. Retching if a patient has already emptied his or her gastric contents is also considered vomiting episode. A distinct episode is characterized by a clear break in vomiting activity of at least 5 minutes
* Emesis must have been nonbloody (streaks of blood presumed due to force of retching are allowed)
* All patients (and a parent or guardian for patients <age 18) must sign informed consent.

Exclusion Criteria:

* Severe dehydration. Severe dehydration is defined as two or more of the following criteria in the presence of decreased intake and increased output due to vomiting or diarrhea: Absent or severely decreased urine output; weak pulse and/or low blood pressure; parched mucous membranes; lethargy, confusion, delirium or loss of consciousness
* Signs and symptoms severe enough to require immediate parenteral hydration and/or parenteral antiemetic medication
* Temperature>39.0
* Likely etiologies for acute vomiting and diarrhea other than acute infectious or toxic gastroenteritis or gastritis. This includes signs of an acute abdomen, which may require surgical intervention
* Chemically-induced gastroenteritis, e.g., from alcohol, other drugs of abuse or other irritant chemicals
* Use within 24 hours of study entry of specific medication for treatment of nausea and/or vomiting, e.g., 5-HT3 antagonists or phenothiazines, or receipt of any IV fluid for any reason. Nonspecific gastrointestinal remedies, such as antacids, proton pump inhibitors and homeopathic remedies, are permitted.
* Congestive heart failure, bradyarrhythmia (baseline pulse<55/min), known long QT syndrome
* Patient who have known QTc prolongation > 450 msec, noted on prior or screening ECG, or who are taking medication known to cause QT prolongation. Note: for current list of medications known to cause QT prolongation see: https://www.crediblemeds.org/healthcare-providers/drug-list/ Use list showing drugs with known risk TdP.
* Known underlying disease which could affect assessment of hydration or modify outcome of treatment, e.g., renal failure, diabetes mellitus, liver disease, alcoholism. Patients with type 2 diet-controlled diabetes mellitus whose baseline blood glucose is <200 may be entered into the study
* Abdominal surgery within the past 3 months
* History of bariatric surgery or bowel obstruction at any time
* Hypersensitivity or other known intolerance to ondansetron or other 5-HT3 antagonists
* Patient has taken apomorphine within 24 hours of screening
* Patient has previously participated in this study
* Patient has participated in another interventional clinical trial, for any indication, in the past 30 days
* For women of childbearing potential: documented or possible pregnancy.

Ages: 12 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2014-12-08 (Actual); Primary Completion 2017-02-13 (Actual); Study Completion 2017-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Silverman, MD, Principal Investigator — Long Island Jewish Hospital (LIJ)
Locations (26):
- United States (26):
  - Kern Medical Center, Bakersfield, California
  - UC Davis, Sacramento, California
  - Olive View- UCLA Medical Center, Sylmar, California
  - George Washington University, Washington D.C., District of Columbia
  - University of Florida Jacksonville, Jacksonville, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - South Shore Hospital, South Weymouth, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Wayne State University - Sinai Grace Hospital, Detroit, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Washington University - St. Louis, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Kings County Hospital, Brooklyn, New York
  - University Hospital of Brooklyn, Brooklyn, New York
  - North Shore University Hospital, Manhasset, New York
  - Cohen's Children's Medical Center of NY, New Hyde Park, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Staten Island University Hospital North, Staten Island, New York
  - Stony Brook University, Stony Brook, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UPMC Mercy, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - CityDoc Urgent Care, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - McAllen Primary Care, McAllen, Texas

REFERENCES:
- [Derived] Silverman RA, House SL, Meltzer AC, Hahn B, Lovato LM, Avarello J, Miller JB, Kalfus IN, Fathi R, Raday G, Plasse TF, Yan EC. Bimodal Release Ondansetron for Acute Gastroenteritis Among Adolescents and Adults: A Randomized Clinical Trial. JAMA Netw Open. 2019 Nov 1;2(11):e1914988. doi: 10.1001/jamanetworkopen.2019.14988. PMID 31702802

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient randomized: 08 December 2014 Last patient completed: 17 February 2017
  This study was conducted in Emergency Departments (EDs) and urgent care centers across the United States. Only 2 sites were urgent care centers; the rest were EDs.
Groups:
- RHB-102: 1 tablet containing 6 mg immediate release and 18 mg sustained release ondansetron, once daily for up to 4 days.
- Placebo: 1 tablet of matching placebo, once daily for up to 4 days.
Period: Overall Study
Arm/Group | RHB-102 | Placebo
Started (ITT Population (treated)) | 192 (6 participants that enrolled in the study did not receive allocated intervention.) | 129 (3 participants that enrolled in the study did not receive allocated intervention.)
Randomized | 198 | 132
Completed | 180 | 118
Not Completed | 12 | 11
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 7 | 5
Not completed — Protocol Violation | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Unkonwn | 1 | 3
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RHB-102 | Placebo | Total
Number analyzed (Participants) | 192 | 129 | 321
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (11.92) | 28.4 (9.69) | 29.0 (11.08)
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 15 | 11 | 26
  18 years or older | 177 | 118 | 295
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122 | 73 | 195
  Male | 70 | 56 | 126
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 1 | 1
  Asian | 13 | 11 | 24
  Black or African American | 80 | 56 | 136
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  White | 77 | 46 | 123
  Other | 21 | 14 | 35
  Hispanic/Latino | 49 | 28 | 77
  Not Hispanic/Latino | 140 | 99 | 239
Nausea [Count of Participants; unit: Participants]
  No nausea | 2 | 3 | 5
  Mild nausea | 24 | 15 | 39
  Moderate nausea | 38 | 40 | 78
  Severe nausea | 70 | 44 | 114
  Nausea as bad as could be | 58 | 27 | 85

OUTCOME MEASURES:

1. Primary Outcome: Treatment Success From 30 Minutes Through 24 Hours After First Dose of Study Medication - ITT Population
Description: Number of patients without further vomiting, without rescue medication, and who were not given intravenous hydration from 30 minutes post first dose until 24 hours post dose
Time Frame: 24 Hours
Population: The Intent-to-treat (ITT) Population consisted of all patients who received any study medication, even if they vomited shortly after administration or were unable to swallow the medication.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo Oral Tablet: 1 tablet of matching placebo, once daily for up to 4 days.
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 192 | 129
Participants
  All ages | 126 | 70
  <18 years of age: number analyzed (Participants) | 15 | 11
  <18 years of age | 12 | 5
  18 years of age or older: number analyzed (Participants) | 177 | 118
  18 years of age or older | 114 | 65
Statistical Analysis 1: Comparison: RHB-102 vs Placebo Oral Tablet; The odds ratio and p-value were from a Cochran-Mantel-Haenszel test. For the 'All ages' category, the odds ratio and p-value were stratified by age; Test type: Superiority; p = 0.0406, Cochran-Mantel-Haenszel — This P-Value is for the "All ages" group; Stratified by age; Odds Ratio (OR) = 1.6081, 95% CI 2-sided [1.0194 to 2.5368]
Statistical Analysis 2: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.0729, Cochran-Mantel-Haenszel — This P-Value is for the "<18 years of age" group; Odds Ratio (OR) = 4.800, 95% CI 2-sided [0.8470 to 27.2024]
Statistical Analysis 3: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.1089, Cochran-Mantel-Haenszel — This P-Value is for the "18 years of age and older" group; Odds Ratio (OR) = 1.4755, 95% CI 2-sided [0.9170 to 2.3741]

2. Secondary Outcome: Responders Through 4 Days After First Dose of Study Medication - ITT Population
Description: Treatment success, as defined in the primary outcome, through 4 days following first dose of study medication.
Time Frame: 4 Days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 192 | 129
Participants | 114 | 67
Statistical Analysis 1: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.1843, Cochran-Mantel-Haenszel; Stratified by age; Odds Ratio (OR) = 1.3545, 95% CI 2-sided [0.8647 to 2.1216]

3. Secondary Outcome: Number of Participants Who Vomited - ITT Population
Description: Analysis of vomiting from 30 minutes after first administration of study medication until 24 hours post first dose
Time Frame: 24 Hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 192 | 129
Participants
  Yes | 38 | 33
  No | 131 | 71
  Missing | 23 | 25
Statistical Analysis 1: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.0166, Cochran-Mantel-Haenszel; Stratified by age; Odds Ratio (OR) = 1.7520, 95% CI 2-sided [1.1058 to 2.7760]

4. Secondary Outcome: Number of Patients Receiving Rescue Antiemetic Therapy - ITT Population
Description: Patients receiving rescue antiemetic therapy within 24 hours after the first dose of study medication.
Time Frame: 24 Hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 192 | 129
Participants | 48 | 43
Statistical Analysis 1: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.1049, Cochran-Mantel-Haenszel; Stratified by age; Odds Ratio (OR) = 0.6677, 95% CI 2-sided [0.4093 to 1.0892]

5. Secondary Outcome: Number of Patients Receiving Intravenous Fluids - ITT Population
Description: Patients receiving parenteral hydration within 24 hours after the first dose of study medication.
Time Frame: 24 Hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 192 | 129
Participants | 34 | 32
Statistical Analysis 1: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.1235, Cochran-Mantel-Haenszel; Stratified by age; Odds Ratio (OR) = 0.6566, 95% CI 2-sided [0.3826 to 1.1268]

6. Secondary Outcome: Severity of Nausea at Baseline - ITT Population
Description: Severity of nausea was assessed using a 5-point Likert scale: 0=no nausea; 1=mild nausea; 2=moderate nausea; 3=severe nausea; 4=nausea as bad as can be.
Time Frame: Day 1 - Baseline through 5 Hours Post Dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 192 | 129
score on a scale
  Baseline | 2.8 (1.03) | 2.6 (1.02)
  Hour 1 Post Dose | 1.1 (1.10) | 1.3 (1.16)
  Hour 2 Post Dose | 0.8 (0.97) | 0.9 (1.07)
  Hour 3 Post Dose | 0.5 (0.85) | 0.8 (1.05)
  Hour 4 Post Dose | 0.4 (0.75) | 0.6 (1.04)
  Hour 5 Post Dose | 0.1 (0.42) | 0.2 (0.49)

7. Secondary Outcome: Incidence and Severity of Diarrhea - ITT Population
Description: Severity of diarrhea for patients having bowel movements was assessed using the Bristol Stool Scale ("BSS"), a Likert scale rating bowel movements from 1=separate hard lumps, like nuts, to 7=watery, no solid pieces; entirely liquid. The BSS was added to the emergency room day and follow-up diaries beginning with protocol amendment 3.
Time Frame: From 30 Minutes Through 24 Hours after First Dose of Study Medication
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 95 | 62
Participants
  No bowel movement | 48 | 29
  BSS 1 | 2 | 2
  BSS 2 | 1 | 2
  BSS 3 | 6 | 2
  BSS 4 | 10 | 5
  BSS 5 | 6 | 2
  BSS 6 | 3 | 7
  BSS 7 | 19 | 13
Statistical Analysis 1: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.5890, Wilcoxon (Mann-Whitney) — This P-Value is for the BSS=7 group

8. Secondary Outcome: Time to Discharge From Emergency Department (ED), Extended Observation Unit, or Hospital - ITT Population
Description: Time from first dose of study medication to discharge from ED, extended observation unit or hospital, whichever comes last, and when clinically appropriate.
Time Frame: Hours from first dose of study medication to discharge from ED, extended observation unit or hospital, whichever comes last
Population: Patients were required to stay in the ED for at least 2 hours (first 172 patients) and subsequently, when post-treatment ECGs were introduced, for 4 hours. Since not all patients had prolonged ED stays, a difference in time until patients were clinically eligible for discharge may have been masked.
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 192 | 129
Hours
  All ages | 4.3 [4.1 to 4.5] | 4.3 [4.0 to 4.6]
  < 18 years of age: number analyzed (Participants) | 15 | 11
  < 18 years of age | 4.3 [2.9 to 4.7] | 4.8 [3.0 to 6.8]
  18 years of age or older: number analyzed (Participants) | 177 | 118
  18 years of age or older | 4.3 [4.1 to 4.5] | 4.2 [4.0 to 4.6]
Statistical Analysis 1: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.8487, Cox proportioanl hazards method — This P-Value is for the "All ages" group; Stratified by age; Hazard Ratio (HR) = 0.9782, 95% CI 2-sided [0.7803 to 1.2264]
Statistical Analysis 2: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.3479, Cox proportional hazards method — This P-Value is for the "<18 years of age" group; Hazard Ratio (HR) = 1.4756, 95% CI 2-sided [0.6549 to 3.3250]
Statistical Analysis 3: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.6332, Cox proportional hazards method — This P-Value is for the "18 years of age of older" group; Hazard Ratio (HR) = 0.9445, 95% CI 2-sided [0.7469 to 1.1943]

9. Secondary Outcome: Time to Resumption of Normal Activities (Work/School/Household) - ITT Population
Description: Time from first dose of study medication to resumption of normal activities (work/school/household).
Time Frame: Hours from first dose of study medication to resumption of normal activities
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Hours
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 192 | 129
Hours
  All ages | 3 [3 to 4] | 3 [3 to 4]
  < 18 years of age: number analyzed (Participants) | 15 | 11
  < 18 years of age | 2 [1 to 4] | 4 [2 to 5]
  18 years of age or older: number analyzed (Participants) | 177 | 118
  18 years of age or older | 3 [3 to 4] | 3 [NA to NA]
Statistical Analysis 1: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.8289, Cox proportional hazards method — This P-Value was for the "All ages" group; Stratified by age; Hazard Ratio (HR) = 1.0275, 95% CI 2-sided [0.8036 to 1.3138]
Statistical Analysis 2: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.3241, Cox proportional hazards method — This P-Value is for the "<18 years of age" group; Hazard Ratio (HR) = 1.5744, 95% CI 2-sided [0.6388 to 3.8802]
Statistical Analysis 3: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.9511, Cox proportional hazards method — This P-Value is for the "18 years of age or older" group; Hazard Ratio (HR) = 0.9920, 95% CI 2-sided [0.7688 to 1.2801]

10. Secondary Outcome: Number of Patients Requiring Hospitalization - ITT Population
Description: Number of patients requiring hospitalization. 4 patients in the RHB-102 treatment group and 1 patient in the placebo treatment group were hospitalized due to lack of efficacy. The remaining patients hospitalized were admitted for reasons other than gastroenteritis.
Time Frame: Day 1 of Study - Day 5 of Study
Population: The number of treated patients requiring hospitalization was low in this study (14 patients). In the RHB-102 group, 11 patients (5.7%) were hospitalized, including one who returned to the ED for gastrointestinal symptoms 2 days after initial treatment. In the placebo treatment group, 3 patients (2.3%) were hospitalized.
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 192 | 129
Participants | 11 | 3
Statistical Analysis 1: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.2005, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.3012, 95% CI 2-sided [0.6221 to 8.5129]

11. Secondary Outcome: Number of Patients Returning to Emergency Department - ITT Population
Description: Proportion of patients returning to emergency department for gastrointestinal symptoms within 4 days of initial discharge
Time Frame: Day 1 of Study - Day 5 of Study
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 192 | 129
Participants | 4 | 4
Statistical Analysis 1: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.5720, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.6674, 95% CI 2-sided [0.1638 to 2.7191]

12. Other Pre Specified Outcome: Treatment Success From 30 Minutes Through 24 Hours After First Dose of Study Medication by Baseline Nausea Severity - ITT Population, All Ages
Description: Proportion of patients without further vomiting, without rescue medication, and who were not given intravenous hydration from 30 minutes post first dose until 24 hours post dose
Time Frame: 24 Hours
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 192 | 129
Participants
  No nausea or mild nausea: number analyzed (Participants) | 26 | 18
  No nausea or mild nausea | 22 | 13
  Moderate nausea: number analyzed (Participants) | 38 | 40
  Moderate nausea | 26 | 24
  Severe nausea: number analyzed (Participants) | 70 | 44
  Severe nausea | 47 | 22
  Nausea as bad as it could have been: number analyzed (Participants) | 58 | 27
  Nausea as bad as it could have been | 31 | 11
Statistical Analysis 1: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.3186, Cochran-Mantel-Haenszel — This P-Value is for the "No nausea or mild nausea" group; Stratified by age; Odds Ratio (OR) = 2.1591, 95% CI 2-sided [0.4770 to 9.7735]
Statistical Analysis 2: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.3473, Cochran-Mantel-Haenszel — This P-Value is for the "Moderate nausea" group; Stratified by age; Odds Ratio (OR) = 1.5750, 95% CI 2-sided [0.6096 to 4.0696]
Statistical Analysis 3: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.0633, Cochran-Mantel-Haenszel — This P-Value is for the "Severe nausea" group; Stratified by age; Odds Ratio (OR) = 2.0971, 95% CI 2-sided [0.9614 to 4.5747]
Statistical Analysis 4: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.2797, Cochran-Mantel-Haenszel — This P-Value is for the "Nausea as bad as it could have been" group; Stratified by age; Odds Ratio (OR) = 1.6397, 95% CI 2-sided [0.6649 to 4.0437]

13. Other Pre Specified Outcome: Treatment Success From 30 Minutes Through 24 Hours After First Dose of Study Medication - PP Population
Description: as for outcome 12
Time Frame: 24 Hours
Population: The Per Protocol Population contained all patients who met all inclusion/exclusion criteria, received a second dose of study medication if they vomited within 15 minutes of receiving the first dose, & did not have a primary diagnosis upon discharge from ED (or, if admitted, discharge from the hospital) other than acute gastroenteritis/gastritis.
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 177 | 122
Participants
  All ages | 123 | 67
  <18 years of age: number analyzed (Participants) | 14 | 11
  <18 years of age | 11 | 5
  18 years of age or older: number analyzed (Participants) | 163 | 111
  18 years of age or older | 112 | 62
Statistical Analysis 1: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.0103, Cochran-Mantel-Haenszel — This P-Value is for the "All ages" group; Stratified by age; Odds Ratio (OR) = 1.8673, 95% CI 2-sided [1.1572 to 3.0131]
Statistical Analysis 2: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.0934, Cochran-Mantel-Haenszel — This P-Value is for the "<18 years of age" group; Odds Ratio (OR) = 4.4000, 95% CI 2-sided [0.7699 to 25.1450]
Statistical Analysis 3: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.0303, Cochran-Mantel-Haenszel — This P-Value is for the "18 years of age or older" group; Odds Ratio (OR) = 1.7356, 95% CI 2-sided [1.0527 to 2.8615]

14. Post Hoc Outcome: Primary Endpoint Subgroup Analysis - PP Population
Description: Examination of treatment success rates by age (<18 and ≥18 years).
Time Frame: 24 Hours
Population: The Per Protocol (PP) Population contained all patients who met all inclusion/exclusion criteria, received a second dose of medication if they vomited within 15 minutes of receiving first dose, and did not have a primary diagnosis upon discharge from the ED (or, if admitted, discharge from the hospital) other than acute gastroenteritis/gastritis.
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 177 | 122
Participants
  < 18 years of age: number analyzed (Participants) | 14 | 11
  < 18 years of age | 11 | 5
  18 years of age or older: number analyzed (Participants) | 163 | 111
  18 years of age or older | 112 | 62
Statistical Analysis 1: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.0924, Cochran-Mantel-Haenszel — This P-Value is for the "<18 years of age" group; Odds Ratio (OR) = 4.4000, 95% CI 2-sided [0.7699 to 25.1450]
Statistical Analysis 2: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.0303, Cochran-Mantel-Haenszel — This P-Value is for the "18 years of age or older" group; Odds Ratio (OR) = 1.7356, 95% CI 2-sided [1.0527 to 2.8615]

15. Post Hoc Outcome: Treatment Success From 30 Minutes Through 24 Hours After First Dose of Study Medication - ITT Population (Logistic Regression Adjusted by Baseline Nausea Severity)
Description: Number of patients without further vomiting, without rescue medication, and who were not given intravenous hydration from 30 minutes post first dose until 24 hours post dose (analyzed using logistic regression with treatment as a factor and baseline nausea severity as a continuous variable)
Time Frame: 24 Hours
Population: The Intent-to-treat (ITT) Population consisted of all patients who received any study medication, even if they vomited shortly after administration or were unable to swallow the medication. The primary efficacy analysis was conducted using the ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 192 | 129
Participants | 126 | 70
Statistical Analysis 1: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.0152, Regression, Logistic; Odds Ratio (OR) = 1.7922, 95% CI 2-sided [1.1188 to 2.8710]

16. Post Hoc Outcome: Treatment Success From 30 Minutes Through 24 Hours After First Dose of Study Medication - PP Population (Logistic Regression Adjusted by Baseline Nausea Severity)
Description: as for outcome 15
Time Frame: 24 Hours
Population: The Per Protocol Population contained all patients who met all inclusion/exclusion criteria, received a second dose of medication if they vomited within 15 minutes of receiving the first dose, and did not have a primary diagnosis upon discharge from the ED (or, if admitted, discharge from the hospital) other than acute gastroenteritis/gastritis.
Measure: Count of Participants; unit: Participants
Arm/Group | RHB-102 | Placebo Oral Tablet
Number analyzed (Participants) | 177 | 122
Participants | 123 | 67
Statistical Analysis 1: Comparison: RHB-102 vs Placebo Oral Tablet; Test type: Superiority; p = 0.0037, Regression, Logistic; Odds Ratio (OR) = 2.0789, 95% CI 2-sided [1.2676 to 3.4095]

ADVERSE EVENTS:
Time Frame: 2 years, 3 months
Description: A treatment-emergent adverse event (TEAE) is an adverse event occurring from the start of study medication.
Arm/Group | RHB-102 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/193 | 0/128
Serious Adverse Events (participants affected / at risk) | 5/193 | 2/128
Other Adverse Events (participants affected / at risk) | 44/193 | 19/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RHB-102 (N=193) | Placebo (N=128)
Bile Duct Stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Sideroblastic Anaemia (Blood and lymphatic system disorders) | 1 | 0
Hospitalization for further diagnosis (Investigations) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 1
Renal Failure Acute (Renal and urinary disorders) | 1 | 0
Diverticulitis Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RHB-102 (N=193) | Placebo (N=128)
Abdominal Distension (Gastrointestinal disorders) | 3 | 1
Abdominal Pain (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 9 | 1
Chest Pain (General disorders) | 2 | 2
Pyrexia (General disorders) | 3 | 5
Dizziness (Nervous system disorders) | 2 | 2
Headache (Nervous system disorders) | 22 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution will provide to Sponsor, for review and comment, all manuscripts or other material prior to such publication. Sponsor shall have 30 days to review any such publication. The Sponsor can require changes to the communication and such confidential information shall be deleted and/or the submission of the proposed publication shall be delayed for an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-06-09): https://cdn.clinicaltrials.gov/large-docs/39/NCT02246439/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-29): https://cdn.clinicaltrials.gov/large-docs/39/NCT02246439/SAP_001.pdf